CLINICAL TRIAL: NCT03220191
Title: A Phase 1, Open-label, 2-period, Fixed Sequence Study Of The Effect Of A Proton Pump Inhibitor On The Relative Bioavailability Of The Proposed Commercial Tablet Formulation Of Palbociclib In Healthy Volunteers
Brief Title: Proton Pump Inhibitor (PPI, Rabeprazole) Effect On Tablet Formulation Of Palbociclib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: A5481091
Record Dates: First submitted 2017-06-16; First posted 2017-07-18 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — palbociclib; Rabeprazole

STUDY DESIGN:
Intervention Model Description: the subjects will receive palbociclib alone in period 1, and receive palbociclib with rabeprazol in period 2
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- palbociclib tablet with/without PPI (Experimental): palbociclib tablet formulation alone in period 1 + palbociclib tablet formulation plus rabeprazole in period 2
  Interventions: Drug: Palbociclib; Drug: Rabeprazole

INTERVENTIONS:
Drug: Palbociclib — palbociclib tablet formulation
  Other Names: Ibrance
Drug: Rabeprazole — rabeprazole as PPI
  Other Names: PPI

SUMMARY:
to evaluate the effect of the PPI (rabeprazole) on the PK of a potential commercial tablet formulation of palbociclib

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment in the study:

1. Healthy female subjects of non childbearing potential and/or male subjects who, at the time of screening, are between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure (BP) and pulse rate (PR) measurement, 12 lead electrocardiogram (ECG) and clinical laboratory tests.

   Female subjects of non childbearing potential must meet at least one of the following criteria:
   1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; status will be confirmed by having a serum follicle stimulating hormone (FSH) level confirming the post menopausal state;
   2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
   3. Have medically confirmed ovarian failure. All other female subjects (including females with tubal ligations) are considered to be of childbearing potential.
2. Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
3. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
4. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

Subjects with any of the following characteristics/conditions will not be included in the study:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Any condition possibly affecting drug absorption (eg, gastrectomy, achlorhydria, peptic ulcer disease).
3. A positive urine drug screen.
4. History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of Screening.
5. Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of study medication (whichever is longer).
6. Screening supine BP >= 140 mm Hg (systolic) or >= 90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is >= 140 mm Hg (systolic) or >= 90 mm Hg (diastolic), the BP should be repeated two more times and the average of the three BP values should be used to determine the subject's eligibility.
7. Screening supine 12 lead ECG demonstrating a corrected QT (QTc) interval >450 msec. If QTc exceeds 450 msec, the ECG should be repeated 2 more times and the average of the 3 QTc values should be used to determine the subject's eligibility.
8. Subjects with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

   * Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) or alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) above the upper limit of normal (ULN).
   * Total bilirubin >= 1.5x ULN; subjects with a history of Gilbert's syndrome may have a direct bilirubin measured and would be eligible for this study provided the direct bilirubin is not greater than 0.5 mg/dL.
9. Pregnant or breastfeeding female subjects; female subjects of childbearing potential; male subjects with partners currently pregnant; male subjects able to father children who are unwilling or unable to use two highly effective methods of contraception as outlined in Section 4.4 of this protocol for the duration of the study and for 90 days after the last dose of investigational product (IP).
10. Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of IP. As an exception, acetaminophen/paracetamol may be used at doses of <= 1 g/day. Limited use of non prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case by case basis following approval by the sponsor.

    Herbal supplements, drugs that increase gastric pH (eg, PPI, H2-receptor antagonist, local antacids), and hormonal contraceptives (including oral and transdermal contraceptives, injectable progesterone, progestin subdermal implants, progesterone-releasing intrauterine devices (IUDs), and postcoital contraceptive methods) and hormone replacement therapy must have been discontinued at least 28 days prior to the first dose of palbociclib.

    Depo Provera must have been discontinued at least 6 months prior to the first dose of palbociclib.
11. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
12. History of sensitivity to heparin or heparin induced thrombocytopenia.
13. History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HepBsAg), hepatitis B core antibody (HepBcAb), or hepatitis C antibody (HCVAb).
14. Use of tobacco or nicotine containing products within 3 months of screening or a positive urine cotinine test (ie, active smokers and those who currently use nicotine containing products are excluded from participation in this study).
15. Unwilling or unable to comply with the Lifestyle guidelines described in this protocol.
16. Subjects who are investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
17. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior, or laboratory abnormality that may increase the risk associated with study participation or IP administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
18. History of known sensitivity to rabeprazole.
19. History of known sensitivity to palbociclib or any of its ingredients.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2017-09-03 (Actual); Study Completion 2017-09-26 (Actual)

PRIMARY OUTCOMES:
AUCinf | PK samples collected from time 0 to 120 hours post-dose
  area under the plasma concentration versus time curve from time 0 to infinity
Cmax | PK samples collected from time 0 to 120 hours post-dose
  maximum plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481091&StudyName=A+Phase+1%2C+Open-label%2C+2-period%2C+Fixed+Sequence+Study+Of+The+Effect+Of+A+Proton+Pump+Inhibitor+On+The+Relative+Bioavailability+Of+The+Proposed+Commercial+Tablet+Formulation+Of+Palbociclib+In+Healthy+Volunteers